CLINICAL TRIAL: NCT04829708
Title: Efficacy and Safety of Prophylactic Cranial Irradiation Versus MRI Surveillance in Patients With Limited-stage Small Cell Lung Cancer Who Achieved Remission After First-line Chemoradiotherapy: a Multicenter Randomized Controlled Phase III Clinical Trial
Brief Title: Efficacy and Safety of Prophylactic Cranial Irradiation Versus MRI Surveillance in Patients With Limited-stage Small Cell Lung Cancer Who Achieved Remission After First-line Chemoradiotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Director of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS-SCLC-III-PCI 2021
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Limited Stage Small Cell Lung Cancer
Keywords: prophylactic cranial irradiation (PCI); MRI surveillance
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI Arm (Active Comparator): Patients received PCI (recommended hippocampal protection) within 6 weeks after first-line treatment, with a total dose of 25 Gy, 2.5 Gy each time, once a day, 5 times a week, a total of 10 times. Brain enhancement MRI examination is performed every 3 months in first two years, and then performed every 6 months until the brain metastasis occur.
  Interventions: Other: MRI Surveillance; Radiation: Prophylactic Cranial Irradiation
- MRI Arm (Experimental): Patients undergo enhancement MRI examination every 3 months in first two years, and then performed every 6 months until the brain metastasis occur. Once brain metastases occur, brain radiotherapy and systemic treatment should be conducted with the follow-up observation of brain enhancement MRI continuing.
  Interventions: Other: MRI Surveillance

INTERVENTIONS:
Other: MRI Surveillance — Receive MRI surveillance
  Other Names: Magnetic Resonance Imaging
Radiation: Prophylactic Cranial Irradiation — Receive PCI
  Other Names: PCI
  Arms: PCI Arm

SUMMARY:
This is a prospective, open,multicenter, randomized controlled phase III clinical trial. In patients with LS-SCLC who achieve remission after first-line chemoradiotherapy, the efficacy and safety of PCI or MRI surveillance is evaluated and analyzed. PCI is performed in hopes of preventing spread of cancer into the brain. The use of brain MRI alone may reduce side effects of receiving PCI and prolong patients' lifespan. MRI surveillance alone (delaying radiation until the actual brain metastasis) may be not inferior to PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of LS-SCLC before first-line chemoradiotherapy (according to the staging system of the Veterans' Affairs Lung Study Group (VALSG), Appendix 2)；
2. Remission is achieved after first-line chemoradiotherapy (CR or PR determined by RECIST v1.1)；
3. Brain MRI examination should be performed to exclude metastatic lesions of brain parenchyma and meninges within four weeks before enrollment；
4. The ECOG PS score was 0~2；
5. The interval between the end of the last treatment cycle and the randomized grouping should be no more than 8 weeks；
6. Estimated survival time ≥ 12 weeks；
7. Patients must agree to participate in the study, comply with the research plan and follow-up process. Written informed consent must obtained.
8. Male or female aged≥18 and≤75 years old;
9. For fertile women and man: Subjects are required to agree to maintain abstinence (no heterosexual intercourse) or use contraception with an annual failure rate of less than 1% during the study treatment period and within at least 6 months after the end of the study treatment period.
10. Hematological indexes: absolute neutrophil count≥1.5×109/ L, platelet count≥75×109 /L, haemoglobin≥9.0g/dL, serum albumin≥3g/dL；
11. Liver function: serum total bilirubin level≤1.5 times normal upper limit (ULN), glutamic pyruvic transaminase, glutamic oxaloacetic transaminase and alkaline phosphatase≤2.5 times ULN；
12. Renal function: defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 15ml/min (Cockcroft-Gault formula, Appendix 4); urinary protein negative or less than 2g in routine urine examination, or 24-hour urinary protein < 1g；
13. Good clotting function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5x ULN;. If the subject is receiving anticoagulant therapy, as long as PT is within the range of anticoagulant use；
14. Women of childbearing age must undergo a urinary pregnancy test within 7 days before the start of treatment and the results are negative and are not breastfeeding.

Exclusion Criteria:

1. Patients with extensive SCLC (Appendix 2)；
2. The subjects are confirmed to have brain or meningeal metastasis before they are randomly divided into groups；
3. During the 5 years before the start of the study, patients with malignant tumors other than SCLC, diseases with negligible risk of metastasis or death (such as expected 5-year OS > 90%) and malignant tumors expected to be cured (such as fully treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated by curable surgery, ductal carcinoma in situ treated by curable surgery)；
4. Previous head and neck radiation fields overlapped with PCI field；
5. MRI examination contraindicated
6. There is evidence that significantly uncontrolled concomitant disease may affect the compliance of the study program, including severe liver disease (such as liver cirrhosis), uncontrollable major seizures or superior vena cava syndrome；
7. Major cardiovascular diseases, myocardial infarction or cerebrovascular events within 3 months before randomization, unstable arrhythmias, or unstable angina pectoris；

   --Patients with known coronary artery disease, congestive heart failure that do not meet the above criteria, or left ventricular ejection fraction ((LVEF)) < 50% must receive a stable treatment plan and optimize it according to the advice of the attending physician, and consult a cardiologist if necessary。
8. Stroke (including hemorrhagic and ischemic) or transient ischemic attack occurred within 6 months before enrollment；
9. There were clinically significant bleeding symptoms or obvious bleeding tendency within 1 month before entering the group, such as gastrointestinal bleeding, gastric ulcer bleeding, active hemoptysis or vasculitis；
10. Serious arteriovenous thrombosis events occurred within 3 months before enrollment, such as deep venous thrombosis, pulmonary embolism, etc. (except for implantable venous infusion port, catheter-derived thrombosis or superficial venous thrombosis, these conditions are not considered "severe" thromboembolism);
11. Diabetic ketoacidosis or hyperglycemia and hyperosmosis occurred in the past 6 months;
12. There was a history of hypertensive crisis and hypertensive encephalopathy;
13. Any other disease, metabolic disorder, abnormal result of physical examination or laboratory examination, and there is reason to suspect that it may affect the reliability of the results of the study or put the patient at high risk of treatment complications；
14. The results of HIV test is positive

    --All patients must be tested for HIV; patients with positive results of HIV will be excluded.
15. Major surgery has been performed within 28 days before the start of the study treatment, or major surgery is expected to be performed during the study period (except those for diagnostic purposes)；
16. Severe infections occur at the beginning of the study, including, but not limited to, infectious complications requiring hospitalization, bacteremia, or severe pneumonia；
17. Pregnant or lactating women；
18. Previous history of severe neurological or mental disorders, including epilepsy, dementia or severe depression that interfere with assessment;
19. The researchers believe that some conditions of the patients may affect the evaluation of the efficacy of this study, as well as the compliance of patients with this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death due to any cause, assessed up to 2 years.
  To compare the efficacy of PCI and MRI surveillance in patients with LS-SCLC.

SECONDARY OUTCOMES:
1-year overall survival rate (1y-OS%) | 1-year
  Rate of patients surviving at 1 year.
3-year overall survival rate (3y-OS%) | 3-year
  Rate of patients surviving at 3 year.
Progression-free survival (PFS) | From the date of randomization until the date of the first onset of disease progression or the time to die of any cause, whichever occurs first, assessed up to 2 years.
Brain metastasis rate | From the date of randomization until the date of occurrence of brain metastasis, assessed up to 2 years.
  To compare brain metastasis rate between the two arms.
Cumulative incidence of neurocognitive impairment | From the date of randomization until the date of occurrence of neurocognitive impairment , assessed up to 2 years.
  To compare the neurocognitive toxicities of PCI and MRI surveillance in patients with LS-SCLC.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (2):
- China (2):
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan

IPD SHARING:
Plan to Share IPD: Undecided